CLINICAL TRIAL: NCT05084872
Title: Hydroxychloroquine in Isolated Cutaneous Mastocytosis Patients or Indolent Systemic Mastocytosis With Associated Skin Involvement Patients: Proof of Concept Study
Brief Title: Hydroxychloroquine in Isolated Cutaneous Mastocytosis Patients or Indolent Systemic Mastocytosis With Associated Skin Involvement Patients
Acronym: HCQMa
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0504; 2020-003268-25 (EudraCT Number)
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Mastocytosis
Keywords: Mastocytosis; mast cell activation symptoms; hydroxychloroquine
MeSH Terms: conditions — Mastocytosis | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will be treated by hydroxychloroquine at a dose of 6 to 6.5mg/kg/day
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Patients will be treated by hydroxychloroquine at a dose of 6 to 6.5mg/kg/day during 12 month

SUMMARY:
The treatment of systemic mastocytosis has two main axes:

* Control of mast cell activation symptoms and
* The control of proliferation (accumulation) of mast cells.

There is no standard treatment and no treatment has a marketing authorization for the treatment of monoclonal indolent mastocytosis.

DETAILED DESCRIPTION:
Mastocytosis is an orphan disease related to the accumulation and / or the proliferation of abnormal mast cells in different tissues.

In adults, a classic distinction is made between isolated cutaneous forms (10 to 15%) and systemic forms (85 to 90%).

The treatment of systemic mastocytosis has two main axes:

* Control of mast cell activation symptoms and
* The control of proliferation (accumulation) of mast cells.

There is no standard treatment and no treatment has a marketing authorization for the treatment of monoclonal indolent mastocytosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Isolated Cutaneous mastocytosis or indolent systemic mastocytosis with associated skin lesions defined according to WHO criteria (and / or international standards for cutaneous mastocytosis)
3. Patient with at least one disability defined by the presence of the following symptoms assessed as moderate to severe:

   1. Cutaneous pruritus with score ≥ 5 on a VAS scale from 0 to 10
   2. Number of flushes / week ≥ 7
4. Skin KIT mutation known
5. Performance scale: OMS/ECOG ≤ 1
6. Woman and man of childbearing age* under effective contraception during all the treatment by hydroxychloroquine, until 8 months after its cessation

Exclusion Criteria:

* Non-symptomatic mastocytosis and / or without skin involvement
* Advanced Systemic mastocytosis
* History of ophthalmic disease and / or cardiac conduction disorders, in particular the prolongation of the QT interval as well as the risk factors for prolongation of the QT interval, such as heart disease (heart failure, myocardial infarction), pro-arrhythmic conditions (eg bradycardia <50 bpm), history of ventricular dysrhythmias, uncorrected hypokalemia and / or hypomagnesemia, concomitant treatment with interval prolonging agents QTagainst-indicating the use of hydroxychloroquine
* Treatment with citalopram, escitalopram, hydroxyzine, domperidone, piperaquine due to the increased risk of ventricular rhythm disorders, especially torsades de pointes
* Specific anti-tumor treatment (chemotherapy, radiotherapy) of less than 4 weeks before inclusion.
* Concomitant specific anti-mast cell treatment
* Contre-indication(s) to XYLOCAINE 10 mg/ml ADRENALINE 0,005 mg/ml, injectable solution: Known hypersensitivity to chlorhydrate de lidocaïne, to amide-type local anaesthetics or one of its excipients (sulfites), patients suffering from recurring porphyrias, coronary insufficiency, ventricular rhythm disorders, severe arterial hypertension, obstructive cardiomyopathy, hyperthyroidism.
* Inclusion in another trial with an experimental therapeutic molecule
* Change symptomatic treatment (including dosage) in the 4 weeks preceding the inclusion visit
* Moderate to severe renal or hepatic failure or diabetes
* History of organ transplant
* Inability to give informed consent
* Inability to undergo medical monitoring for geographical, social or psychic
* Patients with major surgery scheduled in the next two weeks screening
* Patient without health insurance
* Pregnancy, Breastfeeding
* Vulnerable Patient, defined as:
* Esperanzae survival < 6 months
* Patient with another uncontrolled severe disease
* Patient under juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change of mast cell activation symptoms | 12 month
  The primary endpoint of this study is the change of mast cell activation symptoms as pruritus between the start of treatment and 12 months later. Skin pruritus will be assessed by the visual analogue scale from 0 to 10 at each visit.
Change of mast cell activation symptoms | 12 month
  The primary endpoint of this study is the change of mast cell activation symptoms as flushes between the start of treatment and 12 months later. The skin flush will be evaluated according to the absolute number of flushes / week at each visit

SECONDARY OUTCOMES:
Difference on mast cell burden - serum tryptase level | 12 month
  The difference on mast cell burden between the start of treatment and 12 months later will be evaluated by variation of the level serum tryptase l expressed in μg / L.
Difference on skin mast cell burden - mast cells/mm² | 12 month
  The difference on mast cell burden between the start of treatment and 12 months later will be assessed by variation of the number of mast cells / mm² identified on the skin biopsies.
Difference of mast cell activation symptoms : diarrhea | 12 month
  The difference of diarrhea between the start of treatment and 12 months later evaluated by the absolute number of stools / day for diarrhea
Difference of mast cell activation symptoms : pollakiuria | 12 month
  The difference of pollakiuria between the start of treatment and 12 months later assessed by the absolute number of urinations / day for pollakiuria.
Difference of mast cell activation symptoms : arthralgia | 12 month
  The difference of arthralgia between the start of treatment and 12 months later evaluated by the absolute number of painful joints / day and the intensity of joint pain assessed by the visual analogue scale from 0 to 10 for arthralgia.
Difference of mast cell activation symptoms : discomfort | 12 month
  The difference of discomfort between the start of treatment and 12 months later evaluated by the absolute number of faintness / week
The safety of hydroxychloroquine treatment. | 12 month
  The safety of hydroxychloroquine treatment will be done by evaluation of adverse events
effectiveness of treatment | 12 month
  The correlation between the efficacy of treatment with the hydroxychloroquine and level of serum HCQ will be performed by the Bland-Altman test.

CONTACTS AND LOCATIONS:
Overall Officials: Maella Severino-Freire, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Larrey Hospital - Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fradet M, Negretto M, Tournier E, Laurent C, Apoil PA, Evrard S, Degboe Y, Del Mas V, Lamant L, Dubreuil P, Laroche M, Mailhol C, Hermine O, Paul C, Bulai Livideanu C. Frequency of isolated cutaneous involvement in adult mastocytosis: a cohort study. J Eur Acad Dermatol Venereol. 2019 Sep;33(9):1713-1718. doi: 10.1111/jdv.15638. Epub 2019 May 17. PMID 31009132
- [Background] Severino M, Chandesris MO, Barete S, Tournier E, Sans B, Laurent C, Apoil PA, Lamant L, Mailhol C, Laroche M, Fraitag S, Hanssens K, Dubreuil P, Hermine O, Paul C, Bulai Livideanu C. Telangiectasia macularis eruptiva perstans (TMEP): A form of cutaneous mastocytosis with potential systemic involvement. J Am Acad Dermatol. 2016 May;74(5):885-91.e1. doi: 10.1016/j.jaad.2015.10.050. Epub 2016 Feb 19. PMID 26899198